CLINICAL TRIAL: NCT03118388
Title: Engaging Homeless Youth in Vocational Training to Meet Their Mental Health Needs
Acronym: SEI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Kristin Ferguson-Colvin, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34MH082804-01A2 (NIH)
Record Dates: First submitted 2017-04-06; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Mental Disorder; Mental Health; Employment; Housing Problems; Social Support
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being | interventions — Palliative Care; Employment, Supported

STUDY DESIGN:
Intervention Model Description: The SEI model was implemented in four stages: 1) Vocational skill acquisition (4 months); 2) Small business skill acquisition (4 months); 3) SEI formation and product distribution (12 months); and 4) Clinical/case-management services, (ongoing for 20 months). The eight IPS principles were implemented over 20 months by an employment specialist, clinician, and case manager.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 36 SEI youth (Experimental): 36 homeless youth (ages 16-24) randomized to the SEI intervention
  Interventions: Behavioral: Social Enterprise Intervention
- 36 IPS youth (Experimental): 36 homeless youth (ages 16-24) randomized to the IPS intervention
  Interventions: Behavioral: IPS

INTERVENTIONS:
Behavioral: Social Enterprise Intervention — The SEI model was implemented in four stages: 1) Vocational skill acquisition (4 months); 2) Small business skill acquisition (4 months); 3) SEI formation and product distribution (12 months); and 4) Clinical/case-management services, (ongoing for 20 months).
  Other Names: SEI; social enterprise
  Arms: 36 SEI youth
Behavioral: IPS — To implement the IPS at the host agency, one employment specialist, two case managers, and two clinicians were assigned the 22 available IPS cases among them at baseline. Over the 20 months, all IPS participants met individually with the employment specialist, one case manager, and one clinician at least weekly. Regarding job development in the community, the IPS employment specialist also spent about 40% of each week out in the community building relationships with new and existing employers.
  Other Names: Individual Placement and Support; supported employment
  Arms: 36 IPS youth

SUMMARY:
This randomized controlled trial (RCT) compared the efficacy between the Social Enterprise Intervention (SEI) and Individual Placement and Support (IPS) with homeless youth with mental illness.

Methods: Non-probability quota sampling sampling was used to recruit 72 homeless youth from one agency, who were randomized to the SEI (n=36) or IPS (n=36) conditions.

DETAILED DESCRIPTION:
In response to the limited use of RCTs with homeless youth to test research-supported interventions, this study compares the efficacy and short-term outcomes of two interventions that combine employment and clinical services with homeless youth experiencing mental illness. The Social Enterprise Intervention (SEI) is a research-supported intervention using a group approach that engages homeless youth in paid employment as well as case-management and mental health services through involvement in an agency-run social enterprise. The Individual Placement and Support (IPS) model of supported employment is an individually focused, evidence-based intervention , which provides individuals with severe mental illness with customized, long-term, and integrated vocational, case-management, and clinical services to help them gain and maintain competitive employment.

A randomized comparative efficacy trial of the short-term, nonvocational outcomes (depression, self-esteem, social support, housing stability) of the SEI and IPS was conducted over 20 months with 72 homeless youth at a homeless youth drop-in center in Los Angeles. This study answered two research questions: 1) Do homeless youth with mental illness participating in an employment intervention integrated with clinical services (SEI or IPS) experience improvements in their a) mental health status (self-esteem and depression); b) housing stability, and c) social support; and 2) What are the differences between the SEI and IPS groups on mental health, housing stability, and social support outcomes between baseline and follow-up?

ELIGIBILITY:
Inclusion Criteria:

* Age 16-24
* English speaking
* Primary clinical diagnosis in the past year (with at least one symptom in the past 4 weeks) using the DISC-Y interview for one of six mental illnesses (i.e., Major Depressive Episode, Mania/ Hypomania, Generalized Anxiety, Post-traumatic Stress Disorder, Conduct Disorder, and Alcohol/Substance Use Disorders
* Desire to work.

Exclusion Criteria:

* None

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2009-09-18 (Actual); Primary Completion 2011-08-31 (Actual); Study Completion 2011-08-31 (Actual)

PRIMARY OUTCOMES:
Change in depression between baseline and follow-up (using the Adult Self-Report) | 20 months
  Depression was assessed using the Adult Self-Report (ASR) DSM-Oriented Scale for Depressive Problems, consisting of 14 items that measure related emotions and behaviors (Achenbach, 1997). Scoring profiles used normed scales for adults ages 18-35. Higher scores reflected a higher presence of emotions and behaviors. For men, raw scores between 10 and 12 (11 and 13 for women) were within the borderline clinical range, whereas scores 13 and greater (14 and greater for women) were considered in the clinical range.
Change in social support between baseline and follow-up (using the Adult Self-Report) | 20 months
  Social support was a composite-score variable of the sum of four items on the ASR Friends Subscale. The response categories for each item range from none to 5 or more for questions including: "About how many close friends do you have?" The range of scores is from 0 to 12, with higher scores indicating greater social support for the youth.
Change in housing stability status between baseline and follow-up (using a 3-item self-report measure of housing status) | 20 months
  Youth were asked at 20 months about their housing status (i.e., whether they had lived on the streets, in a shelter or institution [i.e., youth or adult shelter, or detention facility, jail, or prison], or in a private residence with family [i.e., biological or foster], relatives, friends, a partner, roommate or alone). Each item was dichotomous and scored as 0 = no or 1 = yes.
Change in self-esteem between baseline and follow-up (using the Rosenberg Self-Esteem Scale) | 20 months
  Self-esteem was measured using the Rosenberg Self-Esteem Scale (RSE; Rosenberg, 1979), a 10-question assessment of feelings about self-worth. Each item is rated using a 4-point Likert-type scale ranging from strongly disagree to strongly agree. Five items are recoded so that higher scores indicate higher levels of self-esteem. The possible range of RSE raw scores is 0 to 30. Scores between 15 and 25 are within normal range, whereas scores below 15 suggest low self-esteem.

IPD SHARING:
Plan to Share IPD: No